CLINICAL TRIAL: NCT03812042
Title: Enzymatic and Genotypic Screening of Lysosomal Storage Diseases in Minority Groups
Brief Title: Screening of Lysosomal Storage Disorders Diseases in Minority Groups
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lysosomal and Rare Disorders Research and Treatment Center, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 16-LDRTC-04
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Lysosomal Storage Diseases
Keywords: Gaucher disease; Fabry disease; Pompe disease; Gangliosidoses
MeSH Terms: conditions — Lysosomal Storage Diseases; Gaucher Disease; Fabry Disease; Glycogen Storage Disease Type II; Gangliosidoses

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screen population: The study population will comprise of patients of healthcare institutions in the Washington, D.C. metro area including but not limited to hospitals, clinics, and doctor's offices.
  Interventions: Diagnostic Test: Enzyme assay and molecular sequencing

INTERVENTIONS:
Diagnostic Test: Enzyme assay and molecular sequencing — Enzyme assay and molecular sequencing on relevant samples conducted from left over blood samples

SUMMARY:
Aim is to undertake a screening study that identifies undiagnosed patients with LSDs and determine the prevalence of these diseases with special focus on underrepresented minority groups.

DETAILED DESCRIPTION:
Lysosomes are small, cytoplasmic organelles that contain several acid hydrolase enzymes. These enzymes break down foreign materials and cellular debris allowing the lysosomes to act as recycling centers for the cells. Following DNA transcription, lysosomal enzymes are produced in the endoplasmic reticulum and targeted to lysosomes by specific recognition markers. If one of the enzymes is absent or if its function is diminished due to either an altered amino acid sequence of the protein or defective intracellular trafficking, the macromolecules metabolized by the specific enzyme will gradually accumulate in the lysosomes. Abnormal substrate storage leads to cellular dysfunction followed by cell death ultimately manifesting as tissue damage and organ failure.

More than 50 metabolic disorders resulting from defective lysosomal enzyme function have been described and are classified as lysosomal storage disorders (LSDs). Although individually uncommon (less than 1 in 100,000), the combined incidence of this group of genetic disorders is about 1 in 5,000 to 1 in 10,000. The prevalence might be even higher than predicted due to undiagnosed instances or misdiagnosis of milder cases.

Most of LSDs are inherited in an autosomal recessive manner except two disorders: Fabry disease and Hunter syndrome, which are X chromosome linked. Two healthy carriers of the same autosomal recessive disease may have an affected child. Usually the carriers are unaware of their carrier status prior to screening or until they have a sick child. These disorders are more common in communities with high consanguinity and where cousin marriages are allowed. In the case of X-linked diseases, the mutant gene is passed down from one generation to the next one in a specific way. If a male has an abnormal copy of the specific gene, he will show the typical presentation of the disease. If a woman has an abnormal copy of the specific gene, she may develop some milder symptoms of the disease due to random X- inactivation.

Screening for LSDs is performed by measuring enzymatic activity in peripheral blood. The most cost effective and convenient way is to use dried filter paper blood spots. A positive screening result has to be followed by a confirmatory enzymatic testing using white blood cells, plasma or cultured skin fibroblasts and/or DNA mutation analysis. The importance of screening for LSDs has been recognized by several state governments as these tests are being included in many newborn screening programs. Although newborn screening helps to identify patients early on, there is still an unmet need for population screening and for identifying patients with reversible tissue damage. LSDs cause serious and progressive problems with multiple body systems. Therapy is available and is promising in most cases. Importantly, patients with LSDs require thorough management plans for their complex health issues.

ELIGIBILITY:
Inclusion Criteria:

* To be enrolled in this study the subject must meet the following (inclusion) criteria:

  * Subject is greater than or equal to 1 day of age and less than or equal to 100 years of age
  * Subject is managed by a physician in the Washington, D.C and Richmond, VA metro area
  * Subject is getting blood work as part of standard clinical care and there is at least 60 uL blood remained in a tube after all clinical tests were run

Exclusion Criteria:

* subjects must not meet any of the following (exclusion) criteria:

  * Absolute contraindication for blood drawing
  * Subject cannot be traced back by the referring physician upon a positive screening result

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise of patients of healthcare institutions in the Washington, D.C. and Richmond, Virginia areas including but not limited to hospitals, clinics, and doctor's offices.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2016-03-17 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Enzyme activity analysis to identify subjects with Lysosomal storage disorders | 5 years
  To identify patients with LSDs using enzymatic activity specific to individual lysosomal storage disorders using left-over blood of blood samples collected as part of standard clinical care.
Genotypic analysis of subjects with abnormal enzyme activity | 5 years
  Samples from subjects with abnormally low enzyme activity will be used for targeted sequencing analysis to diagnose any pathologic mutations.

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Limgala, PhD, Principal Investigator — LDRTC; Margarita M Ivanova, PhD, Principal Investigator — LDRTC; Ozlem Goker-Alpan, MD, Principal Investigator — LDRTC
Locations (1):
- LDRTC, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Institute website for more details — http://www.ldrtc.org